CLINICAL TRIAL: NCT01915368
Title: Determining Optimal Post-Stroke Exercise (DOSE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Janice Eng, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-01933
Record Dates: First submitted 2013-07-11; First posted 2013-08-02 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Cerebrovascular Accident; Stroke; Cerebral Infarction; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases
Keywords: Exercise; Rehabilitation; Dose; Randomized controlled trial; Stroke
MeSH Terms: conditions — Stroke; Cerebral Infarction; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stroke Management Program (SMP) (Active Comparator): Participants will have usual care, and in addition, be provided with periodic information about their progress in the area of mobility using specialized activity monitors
  Interventions: Behavioral: Stroke Management Program (SMP)
- Stroke Monitoring Program (SMonP) (Experimental): Participants will have usual care, and in addition, be progressed according to customized protocols using feedback from specialized activity monitors
  Interventions: Behavioral: Stroke Monitoring Program (SMonP)
- Stroke Supplementary Program (SSP) (Experimental): Participants will have usual care, and in addition, will receive the same as the Stroke Monitoring Group, and also receive one additional hour of daily (5 times per week) physical exercise
  Interventions: Behavioral: Stroke Supplementary Program (SSP)

INTERVENTIONS:
Behavioral: Stroke Management Program (SMP) — Participants will have usual care, and in addition, be provided with periodic information about their progress in the area of mobility using specialized activity monitors
  Arms: Stroke Management Program (SMP)
Behavioral: Stroke Monitoring Program (SMonP) — Participants will have usual care, and in addition, be progressed according to customized protocols using feedback from specialized activity monitors
  Arms: Stroke Monitoring Program (SMonP)
Behavioral: Stroke Supplementary Program (SSP) — Participants will have usual care, and in addition, will receive the same as the Stroke Monitoring Group, and also receive one additional hour of daily (5 times per week) physical exercise
  Arms: Stroke Supplementary Program (SSP)

SUMMARY:
The investigators will conduct a proof-of-concept study to provide preliminary evidence of efficacy of physical exercise dose on ambulatory function in adults undergoing sub-acute stroke rehabilitation.

DETAILED DESCRIPTION:
Participants admitted for stroke rehabilitation will be randomly assigned to either the Stroke Management Group, Stroke Monitoring Group or Stroke Supplementary Group. All three groups will receive usual care, in addition to the intervention. The Stroke Management Group will be provided with periodic information about their progress in the area of mobility using specialized activity monitors. The Stroke Monitoring Group will be progressed according to customized protocols using feedback from specialized activity monitors. The Stroke Supplementary Group will receive the same as the Stroke Monitoring Group, but will also receive one additional hour of daily (5 times per week) physical exercise

ELIGIBILITY:
Inclusion Criteria:

* Have been admitted to a hospital unit for stroke rehabilitation
* Within 10 weeks post-stroke
* 19 years or older
* Are experiencing difficulty walking

Exclusion Criteria:

* Requires greater than one person assist for transfer or ambulation
* Have uncontrolled medical condition or another serious medication condition in addition to stroke
* Unable to understand or follow directions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-09; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Ambulatory function measured by the Six Minute Walk Test | Rehabilitation discharge (average 4-5 weeks post admission)

SECONDARY OUTCOMES:
Ambulatory Function from the Six Minute Walk Test | 6 and 12 months post-stroke
Ambulatory function from the 5 Meter Walk Test | Rehabilitation discharge (average 4-5 weeks post admission) , 6 and 12 months post-stroke
Balance function from the Berg Balance Scale | Rehabilitation discharge (average 4-5 weeks post admission), 6 and 12 months post-stroke
Ambulatory function from the Functional Ambulation Classification | Rehabilitation discharge (average 4-5 weeks post admission), 6 and 12 months post-stroke
Quality of life measured with EuroQol | Rehabilitation discharge (average 4-5 weeks post admission), 6 and 12 months post-stroke
Cognition measured by the Montreal Cognitive Assessment | Rehabilitation discharge (average 4-5 weeks post admission), 6 and 12 months post-stroke
Cognition measured by the Digit Symbols Substitution Test | Rehabilitation discharge (average 4-5 weeks post admission) , 6 and 12 months post-stroke
Cognition measured by the Trail Making Test | Rehabilitation discharge (average 4-5 weeks post admission), 6 and 12 months post-stroke
Depression measured by Patient Health Questionnaire-9 | Rehabilitation discharge (average 4-5 weeks post admission) , 6 and 12 months post-stroke
Heart rate measured during the intervention sessions | From 10 intervention sessions within the 4-week intervention
Step count measured during the intervention sessions | From 10 intervention sessions within the 4-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Janice Eng, PhD, Principal Investigator — The University of British Columbia
Locations (8):
- Canada (8):
  - Fanning Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Laurel Place, Surrey, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - GF Strong Rehab Centre, Vancouver, British Columbia
  - Holy Family Hospital, Vancouver, British Columbia
  - Riverview Health Centre, Winnipeg, Manitoba
  - Toronto Rehabilitation Institute, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ackerley S, Hung SH, Sheehy L, Donkers SJ, Timofeeva P, Best KL, Peters S, Park SS, Ouellet B, Ezeugwu VE, Milot MH, Sakakibara BM, Eng JJ, Connell LA. Exploring factors influencing implementation across the explanatory-to-pragmatic trial continuum: a sequential qualitative integration of delivering higher-intensity walking exercise within inpatient stroke rehabilitation. Implement Sci Commun. 2026 Jan 8. doi: 10.1186/s43058-025-00812-y. Online ahead of print. PMID 41508158
- [Derived] Peters S, Lohse KR, Klassen TD, Liu-Ambrose T, Dukelow SP, Bayley MT, Hill MD, Pooyania S, Yao J, Eng JJ. Higher intensity walking improves global cognition during inpatient rehabilitation: a secondary analysis of a randomized control trial. Front Neurol. 2023 Jun 9;14:1023488. doi: 10.3389/fneur.2023.1023488. eCollection 2023. PMID 37360352
- [Derived] Peters S, Klassen T, Schneeberg A, Dukelow S, Bayley M, Hill M, Pooyania S, Yao J, Eng J. Step Number and Aerobic Minute Exercise Prescription and Progression in Stroke: A Roadmap. Neurorehabil Neural Repair. 2022 Feb;36(2):97-102. doi: 10.1177/15459683211062894. Epub 2021 Dec 23. PMID 34949129
- [Derived] Klassen TD, Dukelow SP, Bayley MT, Benavente O, Hill MD, Krassioukov A, Liu-Ambrose T, Pooyania S, Poulin MJ, Schneeberg A, Yao J, Eng JJ. Higher Doses Improve Walking Recovery During Stroke Inpatient Rehabilitation. Stroke. 2020 Sep;51(9):2639-2648. doi: 10.1161/STROKEAHA.120.029245. Epub 2020 Aug 19. PMID 32811378
- [Derived] Janssen J, Klassen TD, Connell LA, Eng JJ. Factors Influencing the Delivery of Intensive Rehabilitation in Stroke: Patient Perceptions Versus Rehabilitation Therapist Perceptions. Phys Ther. 2020 Feb 7;100(2):307-316. doi: 10.1093/ptj/pzz159. PMID 31711211
- [Derived] Klassen TD, Dukelow SP, Bayley MT, Benavente O, Hill MD, Krassioukov A, Liu-Ambrose T, Pooyania S, Poulin MJ, Yao J, Eng JJ. Determining optimal poststroke exercise: Study protocol for a randomized controlled trial investigating therapeutic intensity and dose on functional recovery during stroke inpatient rehabilitation. Int J Stroke. 2019 Jan;14(1):80-86. doi: 10.1177/1747493018785064. Epub 2018 Jul 16. PMID 30010509
- [Derived] Klassen TD, Semrau JA, Dukelow SP, Bayley MT, Hill MD, Eng JJ. Consumer-Based Physical Activity Monitor as a Practical Way to Measure Walking Intensity During Inpatient Stroke Rehabilitation. Stroke. 2017 Sep;48(9):2614-2617. doi: 10.1161/STROKEAHA.117.018175. Epub 2017 Aug 7. PMID 28784922